CLINICAL TRIAL: NCT05734274
Title: Clinical Effects of Limosilactobacillus Reuteri Probiotics as an Adjunct to the Treatment of Periodontitis: A Randomized Controlled Trial
Brief Title: Clinical Effects of Limosilactobacillus Reuteri Probiotics as an Adjunct to the Treatment of Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, André Marques, Principal investigator - student of the Specialization in Periodontology and Oral Implants, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31/2021
Record Dates: First submitted 2023-01-25; First posted 2023-02-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Periodontitis, Generalized
Keywords: probiotics; Limosilactobacillus reuteri
MeSH Terms: conditions — Chronic Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics Lozenge (Experimental): Subjects are instructed to take a lozenge twice a day, after brushing, in the morning and the evening.
  Interventions: Other: Probiotics
- Negative control Lozenge (Sham Comparator): Subjects are instructed to take a lozenge twice a day, after brushing, in the morning and the evening.
  Interventions: Other: Negative control

INTERVENTIONS:
Other: Probiotics — Probiotics lozenge containing at least 200 million active Limosilactobacillus reuteri.
  Arms: Probiotics Lozenge
Other: Negative control — Sugar-free negative control lozenges.
  Arms: Negative control Lozenge

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of a probiotic lozenge containing Limosilactobacillus reuteri as an adjunct to the periodontal non-surgical treatment of patients with stage II, grade A, B and C, generalized periodontitis.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the effect on disease progression of the probiotic Limosilactobacillus reuteri as an adjunct in the non-surgical periodontal treatment in patients with stage II, grade A, B and C, generalized periodontitis: evaluated by Bleeding on Probing (BoP) - Lindhe, 1972. The secondary purpose is to evaluate the effect of this probiotic on the values of Plaque Index (PI) - Silness & Löe, 1964; Gingival Index (GI) - Löe & Silness, 1963; Probing Pocket Depth (PPD), Clinical Attachment Level (CAL) - Ramfjord, 1959, when compared to a negative control product.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, who intend to voluntarily participate in the study and:

  * Have a definitive diagnosis of stage II, grade A, B or C, generalized periodontitis (2018, World Workshop);
  * Have at least 3 natural teeth maintained per quadrant.

Exclusion Criteria:

* • Patients unable to understand the instructions necessary to participate in the study or unable to give informed consent;

  * Patients who have received any type of periodontal treatment 2 months prior to the start of study participation;
  * Pregnant or breastfeeding patients;
  * Patients with associated systemic pathology, such as diabetes, HIV, asthma, hyperthyroidism, immune system pathologies, lichen erosive or other pathologies treated with corticosteroids or immunosuppressants;
  * Patients undergoing therapy with drugs that may interfere with the response of the gingival tissues: anti-inflammatory drugs, anticonvulsants (phenytoin and sodium valproate), immunosuppressants (cyclosporin-A and tacrolimus) and antihypertensives (nifedipine and verapamil hydrochloride);
  * Patients undergoing anticoagulant therapy;
  * Patients allergic to both lidocaine, articaine and mepivacaine;
  * Patients who require antibiotic prophylaxis for bacterial endocarditis;
  * Patients who have had antibiotic therapy within 2 months of study participation;
  * Patients using chlorhexidine, or other mouthwashes or elixirs;
  * Patients undergoing orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Bleeding on Probing (BoP) - Lindhe, 1972 | 0, 21, 90, 180 days
  Bleeding on probing (in percentage) will be assessed 30 seconds after probing, through a dichotomous scoring system used at six sites per tooth using one (1) and zero (0) for presence or absence, respectively.

SECONDARY OUTCOMES:
Change From Baseline in Plaque Index (PI) - Silness & Löe, 1964 | 0, 21, 90, 180 days
  Each of the four gingival areas of the tooth (mesialbuccal, buccal, distobuccal and palatinal/lingual) is given a score from 0-3; this is the Pl for the area (using plaque discloser. The scores from the four areas of the tooth may be added and divided by four to give the Pl for the tooth. Finally, by adding the indices for the teeth and dividing by the number of teeth examined, the Pl for the individual is obtained.
  Scores criteria:
  0 Absence of microbial plaque.
  1. Thin film of microbial plaque along the free gingival margin.
  2. Moderate accumulation with plaque in the sulcus.
  3. Large amount of plaque in sulcus or pocket along the free gingiva margin.
Change From Baseline in Gingival Index (GI) - Löe e Silness, 1963 | 0, 21, 90, 180 days
  Four gingival areas of the tooth (mesialbuccal, buccal, distobuccal and palatinal/lingual) are given a score from 0 to 3; this is the Gl for the area. The scores from the four areas of the tooth may be added and divided by four to give the GI for the tooth. Finally, by adding the indices for the teeth and dividing by the total number of teeth examined, the Gl for the individual is obtained. The index for the subject is thus an average score for the areas examined.
  Scores criteria:
  0 Normal gingiva: Natural coral pink gingival with no e/o inflammation.
  1. Mild inflammation: Slight changes in color, slight edema. No bleeding on probing.
  2. Moderate inflammation: Redness, edema and glazing. Bleeding upon probing.
  3. Severe inflammation: Marked redness and edema/ulceration/tendency to bleed spontaneously.
Change From Baseline in Probing Depth (PD) | 0, 21, 90, 180 days
  The distance measured from the base of the sulcus or pocket to the free gingival margin.
Change From Baseline in Clinical Attachment Level (CAL) - Ramfjord, 1959 | 0, 21, 90, 180 days
  It is calculated by adding the Probing Pocket Depth to the distance between the cementoenamel junction and the gingival margin (if it is a recession, the value is positive, if it is an increase in gingival volume the recorded value is negative).

CONTACTS AND LOCATIONS:
Overall Officials: André Marques, MDent, Principal Investigator — Estudante da Especialização de Periodontologia e Implantologia
Locations (1):
- Faculty of Dental Medicine - University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei SH, Lang NP. Periodontal epidemiological indices for children and adolescents: II. Evaluation of oral hygiene; III. Clinical applications. Pediatr Dent. 1982 Mar;4(1):64-73. No abstract available. PMID 6960328
- [Background] Montero E, Iniesta M, Rodrigo M, Marin MJ, Figuero E, Herrera D, Sanz M. Clinical and microbiological effects of the adjunctive use of probiotics in the treatment of gingivitis: A randomized controlled clinical trial. J Clin Periodontol. 2017 Jul;44(7):708-716. doi: 10.1111/jcpe.12752. Epub 2017 Jun 23. PMID 28556062
- [Background] Iniesta M, Herrera D, Montero E, Zurbriggen M, Matos AR, Marin MJ, Sanchez-Beltran MC, Llama-Palacio A, Sanz M. Probiotic effects of orally administered Lactobacillus reuteri-containing tablets on the subgingival and salivary microbiota in patients with gingivitis. A randomized clinical trial. J Clin Periodontol. 2012 Aug;39(8):736-44. doi: 10.1111/j.1600-051X.2012.01914.x. Epub 2012 Jun 13. PMID 22694350
- [Background] Vivekananda MR, Vandana KL, Bhat KG. Effect of the probiotic Lactobacilli reuteri (Prodentis) in the management of periodontal disease: a preliminary randomized clinical trial. J Oral Microbiol. 2010 Nov 2;2. doi: 10.3402/jom.v2i0.5344. PMID 21523225
- [Background] Song D, Liu XR. Role of probiotics containing Lactobacillus reuteri in adjunct to scaling and root planing for management of patients with chronic periodontitis: a meta-analysis. Eur Rev Med Pharmacol Sci. 2020 Apr;24(8):4495-4505. doi: 10.26355/eurrev_202004_21032. PMID 32373987
- [Background] Tekce M, Ince G, Gursoy H, Dirikan Ipci S, Cakar G, Kadir T, Yilmaz S. Clinical and microbiological effects of probiotic lozenges in the treatment of chronic periodontitis: a 1-year follow-up study. J Clin Periodontol. 2015 Apr;42(4):363-72. doi: 10.1111/jcpe.12387. Epub 2015 Apr 10. PMID 25728888